CLINICAL TRIAL: NCT05654142
Title: The PIVOT Trial: Project on EHR-Integrated Lifestyle Interventions for Adults Aged Fifty and Older
Acronym: PIVOT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Washington University School of Medicine (Other); University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Jun Ma, MD, PhD, Principal Investigator, Beth and George Vitoux Professor of Medicine, University of Illinois at Chicago
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-1230
Record Dates: First submitted 2022-12-08; First posted 2022-12-16 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: CARDIOMETABOLIC CONDITIONS; Obesity; Pre-diabetes; Metabolic Syndrome; Type2diabetes; Hypertension; Dyslipidemias
MeSH Terms: conditions — Obesity; Glucose Intolerance; Metabolic Syndrome; Hypertension; Dyslipidemias

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group A: Waitlist-Base Intervention (Active Comparator): Participants in Group A will be in the waitlist control condition initially and transition to receive the base intervention at Week 12, which includes 12 GLB video sessions from Week 13-24 and digital messages from Week 25-52.
  Interventions: Behavioral: Base intervention
- Group B: Waitlist-Augmented Intervention (Active Comparator): Participants in Group B will be in the waitlist control condition initially and transition to receive the augmented intervention at Week 12, which includes 12 GLB video sessions plus one-on-one PST from Week 13-24 and digital messages plus group-based PST from Week 25-52. Trained coaches will deliver the PST via videoconference (preferred) or phone.
  Interventions: Behavioral: Augmented Intervention
- Group C: Base Intervention (Responders) (Experimental): Participants in Group C will be the individuals initially randomized to receive the base intervention who achieve 3% weight loss or more by Week 6 after completing the first 6 GLB videos. They will continue the base intervention without re-randomization and complete the next 6 GLB videos from Week 7-12 and receive digital messages from Week 13-52.
  Interventions: Behavioral: Base intervention
- Group D: Base Intervention (Non-responders) (Experimental): Participants in Group D will be the individuals initially randomized to receive the base intervention who do not achieve 3% weight loss by Week 6 after completing the first 6 GLB videos, and who are re-randomized to continue the base intervention. They will complete the next 6 GLB videos from Week 7-12 and receive digital messages from Week 13-52.
  Interventions: Behavioral: Base intervention
- Group E: Augmented Intervention (Non-responders) (Experimental): Participants in Group E will be the individuals initially randomized to receive the base intervention who do not achieve 3% weight loss by Week 6 after completing the first 6 GLB videos, and who are re-randomized to receive the augmented intervention. They will complete the next 6 GLB videos from Week 7-12 and receive digital messages from Week 13-52. They will also work with a trained coach via videoconference (preferred) or phone to receive one-on-one PST from Week 7-24 and group-based PST from Week 25-52.
  Interventions: Behavioral: Augmented Intervention

INTERVENTIONS:
Behavioral: Base intervention — 12 Group Lifestyle Balance videos and digital motivational messages
  Arms: Group A: Waitlist-Base Intervention; Group C: Base Intervention (Responders); Group D: Base Intervention (Non-responders)
Behavioral: Augmented Intervention — 12 Group Lifestyle Balance videos and digital motivational messages plus remote coaching for one-on-one and group-based problem-solving treatment via videoconference (preferred) or phone
  Arms: Group B: Waitlist-Augmented Intervention; Group E: Augmented Intervention (Non-responders)

SUMMARY:
This is a multisite clinical trial of healthy lifestyle programs for middle-to-older-aged adults (50 -74 years) to improve their weight and, therefore, reduce risk for chronic disease. This study will investigate whether a proven, self-directed video-based lifestyle program can be significantly enhanced with the assistance of a coach via videoconference or phone to help people as they adopt healthy eating and exercise behaviors. Additionally, the study will examine what factors might explain why some people achieve better outcomes than others. Understanding this can help to tailor the program to an individual for personalized care in the future.

Importantly, this study aims to demonstrate how readily a digital lifestyle program, with or without remote coaching, can be seamlessly delivered to patients at home via the patient portal of their electronic health record. This practical use of existing telehealth tools could be a feasible and effective means to offer behavioral treatments during routine medical care.

DETAILED DESCRIPTION:
This multisite clinical trial uses a 2-stage sequential randomization design to test the adaptive and nonadaptive augmentation of a validated Group Lifestyle Balance (GLB) video program (base intervention) using problem solving treatment (PST), a proven behavior therapy. The GLB video program will be delivered via the patient portal of the electronic health record system. Trained coaches will deliver PST remotely via videoconference or phone.

English-speaking adults (N=1029), 50-74 years of age with a body mass index ≥27 and ≥1 cardiometabolic conditions, will be randomized at baseline to base intervention or waitlist control. Participants initially randomized to the waitlist control will be re-randomized after a 12-week control period to receive the base (Group A) or the augmented intervention (Group B), without tailoring based on early weight loss. Among participants initially randomized to the base intervention, responders defined by ≥3% weight loss at 6 weeks will continue the base intervention (Group C); nonresponders who are participants with <3% weight loss or missing weight data by 6 weeks will be re-randomized to continue the base intervention alone (Group D) or augmented with PST coaching via videoconference (Group E).

We hypothesize: (1) the augmented intervention will be more effective than the base intervention both among early nonresponders to the base intervention (adaptive) and among participants in the waitlist control condition (nonadaptive) at 52 weeks; (2) the adaptive augmented intervention will be more efficacious than the base intervention and more efficacious than the waitlist control condition at 12 weeks. Aim 2 is to identify predictors of clinically significant (5%) weight loss for individual patients, using sociodemographic, clinical and behavioral engagement characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 - 74 years (inclusive)
* Confirmed body mass index (BMI) ≥27.0 based on:

  * Weight measured by participant at home using the study-provided wireless weight scale
  * Height documented in the EHR during at least 2 separate ambulatory care encounters within the past 2 years
* Diagnosis of 1 or more cardiometabolic condition (prediabetes, metabolic syndrome, type 2 diabetes, hypertension, dyslipidemia) in the EHR
* Willing and able to accept randomization, and provide written informed consent and HIPAA authorization
* Willing and able to participate in all aspects of the data collection and intervention protocols, including remote monitoring with a study-provided wireless weight scale and activity tracker and the use of a study tablet for access of MyChart, REDCap, and Fitbit apps

Exclusion Criteria:

* Unable to speak, read, understand English sufficiently for informed consent
* No reliable Wi-Fi Internet access at home
* Self-report of current active weight loss treatment, including research-based commercial weight loss programs (e.g., Weight Watchers, Jenny Craig, HMR, Omada, TOPS), other weight loss or related behavioral health or wellness programs led by trained personnel (professional or lay) at the recruiting clinic or in the local community, and prescription weight loss medications
* Screen positive for active eating disorder (bulimia nervosa or binge eating disorder) using PHQ- eating disorder module
* Planned or prior bariatric surgery within the last 2 years (Note: patients who are more than 2 years post bariatric surgery can participate if otherwise eligible)
* Unable to pass the Revised Physical Activity Readiness Questionnaire (PAR-Q) or obtain physician medical clearance to participate
* Presence of any significant safety concerns or contraindications related to serious physical or mental health issues based on the EHR or self-report (e.g., type 1 diabetes or insulin dependence, myocardial infarction, stroke, cancer diagnosis (other than non-melanoma skin cancer) within the past 12 months and/or actively receiving cancer treatment, end-stage organ failure, bipolar disorder, psychosis, life expectancy <12 months)
* Cognitive impairment based on the Callahan 6-item screener
* Active alcohol or substance use disorder (including prescription drugs) based on the CAGE Questionnaire Adapted to Include Drugs (CAGE-AID)
* Discontinued health care at the recruiting site, or plan to discontinue in the next 12 months
* Participation in other behavioral, medical or surgical treatment studies by self-report that conflict with the primary weight loss outcome of this study.
* Family/household member of an already enrolled participant or of a study team member
* Investigator discretion for clinical safety or protocol adherence reasons

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1029 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Assess change in weight from baseline to 52 weeks | Baseline, 52 weeks
  All participants will be provided a Fitbit Aria weight scale, a Fitbit Inspire 3 activity tracker, and a study tablet (Samsung Galaxy). At baseline (0) and 52 weeks, a study coordinator at each site who is blinded to randomization will proactively contact participants by phone, email, and/or text to remind them to weigh themselves at the same time on at least 3 days during the week. Participants will be instructed to weigh themselves on their study-provided Aria scale right after waking up and emptying their bladder (and bowel, if possible). They should wear only a t-shirt and undergarments, and bare feet. We will obtain participants' self-monitored weight data using a developed program for automated daily synchronization via the Fitbit open API.

SECONDARY OUTCOMES:
Assess change in weight from baseline to 12 weeks | Baseline, 12 weeks,
  All participants will be provided a Fitbit Aria weight scale, a Fitbit Inspire 3 activity tracker, and a study tablet (Samsung Galaxy). At baseline (0) and 12 weeks, a study coordinator at each site who is blinded to randomization will proactively contact participants by phone, email, and/or text to remind them to weigh themselves at the same time on at least 3 days during the week. Participants will be instructed to weigh themselves on their study-provided Aria scale right after waking up and emptying their bladder (and bowel, if possible). They should wear only a t-shirt and undergarments, and bare feet. We will obtain participants' self-monitored weight data using a developed program for automated daily synchronization via the Fitbit open API.
Assess trajectories of weight change from baseline to 6, 12, 24, and 52 weeks | Baseline, 6 weeks, 12 weeks, 24 weeks
  All participants will be provided a Fitbit Aria weight scale, a Fitbit Inspire 3 activity tracker, and a study tablet (Samsung Galaxy). At baseline (0), 6, 12, 24, and 52 weeks, a study coordinator at each site who is blinded to randomization will proactively contact participants by phone, email, and/or text to remind them to weigh themselves at the same time on at least 3 days during the week. Participants will be instructed to weigh themselves on their study-provided Aria scale right after waking up and emptying their bladder (and bowel, if possible). They should wear only a t-shirt and undergarments, and bare feet. We will obtain participants' self-monitored weight data using a developed program for automated daily synchronization via the Fitbit open API.
Assess changes in number of steps using Fitbit activity tracker at 6, 12, 24 and 52 weeks | Baseline, 6 weeks, 12 weeks, 24 weeks, 52 weeks
  All participants will receive a study-provided Fitbit Inspire 3 activity tracker with heart rate and sleep monitor, assistance with account and device setup. At 0, 6, 12, 24 and 52 weeks, a study coordinator at each site who is blinded to randomization will proactively contact participants by phone, email, and/or text to remind them to wear their activity tracker for at least 10 hours on 3 or more days during the week. We will obtain participants' self-monitored number of steps using a developed program for automated daily synchronization via the Fitbit open API.
Assess changes in physical activity using the International Physical Activity Questionnaire at 6, 12, 24 and 52 weeks | Baseline, 6 weeks, 12 weeks, 24 weeks, 52 weeks
  All participants will self-administer the International Physical Activity Questionnaire (IPAQ), a 7-item questionnaire that captures a participant's physical activity over the last 7 days.
Assess changes in fruit/veggie/fat/fiber intake at 6, 12, 24 and 52 weeks | Baseline, 6 weeks, 12 weeks, 24 weeks, 52 weeks
  Dietary intake will be measured using 17-item fruit, vegetable, fat, and fiber screener by self-report. Correlations between screener estimates and estimated true intake were 0.5-0.8.
Assess changes in efficacy in weight control at 6, 12, 24 and 52 weeks | Baseline, 6 weeks, 12 weeks, 24 weeks, 52 weeks
  Participants will complete validated self-administered scale of self-efficacy for weight control using the Weight Efficacy Lifestyle Questionnaire. Sum of scores of 8 items, with a range between 0 and 80. Higher scores indicate higher self-efficacy to control eating behaviors.
Assess changes in efficacy in diet change at 6, 12, 24 and 52 weeks | Baseline, 6 weeks, 12 weeks, 24 weeks, 52 weeks
  Participants will complete validated self-administered scale of self-efficacy for dietary change using the Eating Habits Confidence Survey. The total score is mean item scores, with a range between 1 and 5. Higher scores indicate higher diet self-efficacy (i.e., higher ability to avoid eating certain unhealthy foods).
Assess changes in efficacy in physical activity at 6, 12, 24 and 52 weeks | Baseline, 6 weeks, 12 weeks, 24 weeks, 52 weeks
  Participants will complete validated self-administered scale of self-efficacy for physical activity using the Exercise Confidence Survey. The total score is mean item scores, with a range between 1 and 5. Higher scores indicate higher exercise self-efficacy (i.e., greater confidence in performing certain behaviors consistently for at least 6 months).
Assess changes in social support/autonomous support per Health Care Climate Questionnaire at 6, 12, 24 and 52 weeks | Baseline, 6 weeks, 12 weeks, 24 weeks, 52 weeks
  Participants will complete the Health Care Climate Questionnaire (HCCQ), which assessed their perceptions of the autonomy supportiveness of their care team. HCCQ contains 15 items, rated on a 5-point scale ranging from "not true at all" to "very true." After reversing the score of a negative item, an average score is calculated with higher score indicating a higher level of perceived autonomy support.
Assess changes in problem solving ability at 6, 12, 24 and 52 weeks | Baseline, 6 weeks, 12 weeks, 24 weeks, 52 weeks
  Participants' problem solving abilities will be assessed using the reliable and valid SPSI-R:S that contains 25 items in the following 5 subscales: positive problem orientation (PPO), negative problem orientation (NPO), rational problem solving (RPS), impulsive/careless style (ICS), and avoidance style (AS). Each item is rated on a 5-point scale ranging from "not at all true of me" (0) to "extremely true of me" (4). SPSI-R:S is a short version of the long SPSI-R:L form which has Cronbach's alpha coefficient of 0.95 for the total score and of 0.67-0.92 for subscales.
Assess changes in patient activation at 6, 12, 24 and 52 weeks | Baseline, 6 weeks, 12 weeks, 24 weeks, 52 weeks
  The 13-item PAM measures patient's self-reported knowledge, skill, and confidence for self-managing his or her health condition. It demonstrated acceptable internal consistency (Conbrach's alpha = 0.81). The 13-item PAM score accounts for 92% of the variation in the activity measured by the original 22-item PAM. The score is also significantly correlated with general preventive behaviors and disease-specific self-management behaviors.
Assess changes in perceived stress at 6, 12, 24 and 52 weeks | Baseline, 6 weeks, 12 weeks, 24 weeks, 52 weeks
  Perceived Stress Scale (PSS) measures the perception of stress (i.e., the degree to which situations in one's life are appraised as stressful). PSS contains 14 items, rated on a 5-point scale ranging from "never" to "very often." After reversing the scores on 7 positive items, a sum of score is calculated with higher score indicating higher perceived stress. Cronbach's alpha ranged from 0.84 to 0.86.
Assess changes in health-related quality of life at 6, 12, 24 and 52 weeks | Baseline, 6 weeks, 12 weeks, 24 weeks, 52 weeks
  The SF-8 is an 8-item version of the SF-36 that measures overall health-related quality of life. Physical and mental health composite scores are computed using the scores of 8 questions and range from 0 to 100, with 0 indicating the lowest level of health and 100 indicating the highest level of health. Correlation between the SF-8 and the SF-36 is 0.825 for physical health component and 0.881 for mental health component.
Assess changes in sleep disturbance score at 6, 12, 24 and 52 weeks | Baseline, 6 weeks, 12 weeks, 24 weeks, 52 weeks
  Sleep disturbance is assessed on the 8-item PROMIS sleep disturbance scale short form which measures symptoms of insomnia. Each item is scaled from 1 (not at all) to 5 (very much). Sleep disturbance score=(Raw sum ×number of items on the short form) / number of items answered. The higher the score the greater sleep disturbance.
Assess changes in sleep impairment score at 6, 12, 24 and 52 weeks | Baseline, 6 weeks, 12 weeks, 24 weeks, 52 weeks
  Sleep impairment is assessed on the 8-item PROMIS sleep-related impairment scale short form which measures symptoms of daytime sleepiness. Each item is scaled from 1 (not at all) to 5 (very much). Sleep impairment score=(Raw sum ×number of items on the short form) / number of items answered. The higher the score the greater sleep impairment.
Assess changes in cognitive functioning at 6, 12, 24 and 52 weeks | Baseline, 6 weeks, 12 weeks, 24 weeks, 52 weeks
  Cognitive functioning will be assessed on the PROMIS version 1.0 short-form subscales of Cognitive Abilities and Cognitive Concerns. Each subscale contains 8 items. The Cognitive Abilities items target positive self-assessments of cognitive functioning such as "My memory has been as good as usual" and "I have been able to concentrate." The Cognitive Concerns items are worded negatively and express concerns in the same areas, for examples, "My thinking has been slow" and "I have had trouble shifting back and forth between different activities that require thinking." Items on both subscales use a 5-point rating from "not at all" to "very much." Items are summed to create a total score for each subscale.
Assess changes in cardiovascular risk at 52 weeks | Baseline, 52 weeks
  The non-laboratory Framingham risk prediction model estimates individuals' 10-year risk of developing any major atherosclerotic cardiovascular disease (CVD) event. The component risk factors are age, BMI, systolic blood pressure, smoking status, presence of diabetes, and medication for high blood pressure. Participants will be asked to confirm their age and report their smoking history at baseline and current smoking status at baseline and 52 weeks. The BMI will be calculated based on participants' self-measured weight data as described above and height measurements abstracted from their EHR. Blood pressure, diagnosis of diabetes, and prescriptions for high blood pressures will also be abstracted from the EHR.
Assess changes in number/severity of comorbidity at 52 weeks | Baseline, 52 weeks
  The Cumulative Illness Rating Scale (CIRS) is a composite index of the number and severity of medical problems by organ system. It has been validated in diverse populations and settings, including primary care patients, with published guidelines and electronic tools for application and scoring using electronic health record (EHR) data.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Department of Medicine, Vitoux Program on Aging and Prevention, Chicago, Illinois
  - Washington University School of Medicine in St Louis, St Louis, Missouri
  - University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania